CLINICAL TRIAL: NCT07023198
Title: Implementing Provider Initiated Clinical Breast Examination and Navigation Intervention to Improve Timely Diagnosis and Initiation of Breast Cancer Treatment at General Hospitals in Ethiopia: A Study Protocol for Implementation Mapping Study
Brief Title: Improving Timely Diagnosis and Initiation of Breast Cancer Treatment in Ethiopia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Addis Ababa University (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Aragaw Tesfaw, Assistant professor, Addis Ababa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Protocol No.034/24/SPH; 81301031 (Other Grant/Funding Number: Research Networks for Health Innovations in Sub-Saharan Africa (RHISSA), NORA)
Record Dates: First submitted 2025-06-05; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; Patient navigation; implementation research; Ethiopia
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: An implementation mapping study will be conducted which is a process framework that provides a systematic, five-step approach to select and evaluate implementation strategies to bring an evidence-based intervention. This design includes: 1) conducting a needs assessment, (2) identify adoption and implementation outcomes, performance objectives, performance determinants, and change objectives), (3) select & design implementation strategies, (4) produce implementation protocols and materials and (5) evaluate implementation outcomes (1). The RE-AIM framework will also be used to evaluate the implementation process and outcome. It is a comprehensive model designed to evaluate and enhance the impact of health interventions, by considering individual and organizational factors that influence the success of health interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical breast examination and navigation (Experimental): Nurses will be trained on clinical breast examination techniques and navigation to routinely offer CBE to eligible women and to support women with suspicious findings until compilation of diagnosis and Initiation of breast cancer treatment
  Interventions: Other: Clinical breast examination and Navigation

INTERVENTIONS:
Other: Clinical breast examination and Navigation — trained nurses on clinical breast examination and navigation will provide screening for all eligible women and they will follow those women who will have suspicious breast lesions until they have completed their final diagnosis of breast cancer and initiation of breast cancer treatment

SUMMARY:
Brief summery Prolonged presentation, along with diagnostic and treatment delays, remain significant problems for breast cancer care in Ethiopia, primarily due to low health-seeking behaviour, lack of access, long waiting times, and weak referral systems. Despite these challenges, evidence-based interventions like structured breast screening and patient navigation services are limited. To address these issues, the investigators aimed to implement a provider-initiated clinical breast examination and patient navigation intervention using an implementation mapping approach.

This is just a one-year implementation mapping (IM) study that will be carried out at four general hospitals in Ethiopia after identifying contextual barriers and implementation determinants using a baseline assessment. The main aim of the study is to improve timely diagnosis and initiation of breast cancer treatment by implementing provider-initiated clinical breast examination and patient navigation interventions.

The study has the following key outcomes: Proportion of CBE uptake, Time to diagnosis, Proportion of early-stage disease, Time to treatment initiation, Barriers and facilitators to implementation, Patient satisfaction, and perceived quality of care The study will strictly follow the steps of implementation mapping design to select and evaluate implementation strategies to bring an evidence-based intervention. In addition, the study will apply established frameworks such as the CFIR and RE-AIM, which can strengthen the study's ability to identify, measure, and interpret multiple implementation outcomes. This study aligns with the Ministry of Health priorities aimed at scaling up breast cancer early detection in general hospitals, which are potential sites for expanding and decentralizing peripheral cancer care in Ethiopia. Therefore, it will provide evidence-based strategies that can be incorporated into the routine health care practice to address multiple points of delay in the care pathway, mainly in the early detection and referral phases at each level of the health care system in the country. The findings will offer a promising strategy to address critical delays in the breast cancer care continuum for low-income settings facing similar challenges. Moreover, the findings will contribute to national and global efforts to improve breast cancer care equity and outcomes through implementation science.

DETAILED DESCRIPTION:
The majority of breast cancer patients experienced long delays from their initial presentation to final diagnosis and treatment initiation in Ethiopia, primarily due to low health-seeking behavior, lack of access, long waiting times for diagnostic workups, and weak referral systems. Despite these challenges, evidence-based interventions like structured breast screening using clinical breast exams and PN services are limited. CBE is offered only for those presenting with breast complaints. Standard screening tools such as mammography are very limited in the country. This urges an urgent need for context-specific implementation strategies that are evidence-based and feasible within the constraints of the health care facilities in Ethiopia, where patients suffer long diagnostic and treatment delays.

The investigators hypothesized that implementing provider-initiated (CBE) and PN would improve the screening uptake, timely diagnosis, and linkage to treatment for breast cancer at general hospitals in Ethiopia. The intervention will be implemented based on the recently launched national breast health guideline, which recommends using CBE and PN services with effective referral pathways. This combined approach aligns with the WHO's GBCI, aiming to reduce mortality through early detection and comprehensive care, and is particularly suited to Ethiopia.

The investigators aimed to use the Implementation Mapping framework, a systematic, step-by-step methodology used to guide the development of implementation strategies that enhance the adoption, execution, and sustainability of evidence-based interventions by engaging stakeholders within local settings. This study will address a critical gap in breast cancer care in Ethiopia by facilitating early detection, timely diagnosis, and care. Moreover, the findings will generate practical insights and scalable approaches that can inform policymakers and be expanded nationally by integrating them into the conventional healthcare system and tailoring them for other low-resource settings facing comparable issues.

Implementation process Our implementation will follow the following five steps of implementation mapping design Step 1: Conduct a needs assessment The first step is conducting a thorough assessment using the CFIR framework to gather general information on the health care infrastructure and workforce, opportunities, and challenges from the perspectives of stakeholders by conducting initial health facility surveys, IDIs, and FGDs.

Step 2: Identify adoption and implementation outcomes, performance objectives, performance determinants, and change objectives In this step, the investigators will identify the potential adoption and implementation outcomes, performance objectives, performance determinants, and change objectives based on our formative assessment findings Step 3: Select and Design Implementation Strategies

In the third step, the investigators identified the following key implementation strategies that address the specific needs of receivers and implementers within the local context:

1. Training healthcare providers in CBE and PN; the investigators will provide comprehensive training for HCPs on CBE and PN using practical demonstrations and role-playing scenarios to enhance their knowledge and skills.
2. Integrating the initiative into routine clinical workflows: the clinical staff working in the hospitals will be oriented to link eligible women to navigators& those who present with breast complaints to the trained breast nurses for CBE & navigation service. We will make all the eligibility criteria and educational materials accessible to all clinical staff and ensure that the initiative becomes a routine part of care.
3. Provider engagement and incentives; Incentive mechanisms that encourage participation in training and the adoption of CBE & PN practices will be developed. This includes recognition awards, professional development opportunities, and financial incentives based on performance metrics.
4. Community engagement and awareness; the investigators will develop awareness creation programs within the hospitals (Morning health education in waiting areas) and community settings using posters, brochures, and social media to educate the public about the importance of breast cancer screening and early detection. Breast cancer survivors, community HEWs, and key informants will be involved to advocate for breast health and screening.
5. Intervention delivery: The navigators will identify eligible women for CBE on each day among the hospital attendants and invite them to undergo a CBE screening at the surgical referral clinic (SRC) with the help of the surgeon. Clinical staff will also identify eligible women from their daily contacts and advice, and link women to the trained nurse for CBE screening. The screening will be held every day at each site. A screening card will be given to the screened women with the date of last screening and the date when the next screening will be. The navigators will have direct communication with clinical staff daily. Navigators will contact referred patients by phone within 2 days of referral, collect baseline data, provide counselling on follow-up and undergoing further evaluation, give date for follow-up within 14 days of referral, send SMS reminder to patient 3 and 1 days before scheduled follow-up, follow-up on whether patient presented for first evaluation at diagnostic center, follow-up 45 days post-referral to check whether patient has completed all recommended testing, keep records of patients' progress until evaluation of breast (confirmed diagnosis) is complete. The navigator will have communications with the referral center to assist her until she finishes all the diagnoses. Local community HEWs will be used to trace women in case access by phone is difficult. The Redcap database will be used to track patient progress and to generate reports that support navigators' and screener's workflow.
6. Monitoring and Feedback: A structured follow-up tool will be developed to track key performance indicators (KPIs) such as the number of CBEs performed, referrals made, and time to diagnosis recorded through the RedCap database. The supervisory team will hold weekly meetings with the providers and monthly onsite supervisions to monitor the progress and ensure adherence to the protocol. Daily feedback will be provided to providers on their performance to encourage continuous improvement.
7. Collaboration with stakeholders; stakeholders at local and national levels, including the regional and MOH officials, local NGOs, hospital leaders, patients, HEWs, and research and academic institutions, will be involved.
8. Addressing barriers to care; a dedicated healthcare professional (trained breast nurses) will be assigned to identify barriers and to guide patients through the healthcare system
9. Sustainability planning; the intervention is being implemented according to the newly launched national breast health guideline recommendations. Ongoing training and support for providers will be planned for the long-term integration of the intervention into routine practice.

Step 4: Produce Implementation Protocols and Materials. In this step, a set of necessary protocols & materials will be developed. This includes health education materials (audio visuals, posters, brochures), follow-up data collection tools, registration log books, screening tickets, HCP training manuals, CBE and PN SOPs, consent forms, patient navigation tracking forms, referral logbooks, post-intervention assessment tools, observation checklists, monitoring and evaluation tools.

Step 5: Evaluation of implementation outcomes In this step, a RE-AIM framework will be used to evaluate the impact of the intervention on improving each of the adoption and implementation outcomes. Surveys and interviews will be conducted with HCPs and patients to understand their perceptions and experiences with the intervention using each domain of the RE-AIM framework.

ELIGIBILITY:
Inclusion Criteria:

* Women aged≥30 years old and presenting to the study hospitals, including attendants, women presenting for various health services, such as outpatient care, maternal and child health services, or other health needs
* Women presented to the general hospitals with any breast abnormalities
* Women with suspicious breast lesions who will be referred from primary health facilities to general hospitals

Exclusion Criteria:

* Women screened for breast cancer in the past year

  * Women who have been treated for breast cancer in the past year and males will be excluded

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis of a suspicious breast lesion | 12 month
  Time from first presentation to confirmed diagnosis of suspicious breast lesion. If < 60 days, it is considered a short interval and if ≥ 60 days, it is considered as long interval
Proportion of clinical breast examination (CBE) uptake | 12 month
  This the percentage of women who undergo CBE from the total eligible women who come to the study hospitals each working day

SECONDARY OUTCOMES:
proportion of early stage diagnosis among suspecious breast lesions | 12 month
  This is the proportion of early-stage disease among total suspicious breast lesions identified. Tumors will be categorized according to the American Joint Committee on Cancer staging manual, 7th edition. All clinical, investigative, and intraoperative findings will be used to stage the disease. Stage 1 (T1N0); stage 2 (IIA=T0N1, T1N1 &T2N0, IIB= T2N1& T3N0,) and stage 3 (IIIA=T0N2, T1N2, T2N2, T3N1&T3N2, IIIB=T4N0, T4N1, T4N2, IIIC= Any T N3) and stage 4 (any T any N and M1). Stage III and IV disease will be defined as 'late stages', and stage I and II disease will be defined as 'early stage' disease
Time to treatment initiation | 12 month
  The time from pathological diagnosis to initiation of the first breast cancer treatment if < 30 days, it is considered as short interval and if ≥30 days, it is considered as long interval

CONTACTS AND LOCATIONS:
Locations (1):
- Butajira, Saint Lukas, Bishoftu, and Halaba kulito hospitals, Addis Ababa, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The data for this study will be shared based on a reasonable request to the principal investigator of the study
Supporting Information: Study Protocol, SAP
Time Frame: From June 7, 2025, to March 23, 2026
Access Criteria: The data in this study are available from the principal investigator upon reasonable request.

REFERENCES:
- [Background] Pace LE, Dusengimana JV, Keating NL, Hategekimana V, Rugema V, Bigirimana JB, Costas-Chavarri A, Umwizera A, Park PH, Shulman LN, Mpunga T. Impact of Breast Cancer Early Detection Training on Rwandan Health Workers' Knowledge and Skills. J Glob Oncol. 2018 Sep;4:1-10. doi: 10.1200/JGO.17.00098. PMID 30241228
- [Background] Hoffman HJ, LaVerda NL, Young HA, Levine PH, Alexander LM, Brem R, Caicedo L, Eng-Wong J, Frederick W, Funderburk W, Huerta E, Swain S, Patierno SR. Patient navigation significantly reduces delays in breast cancer diagnosis in the District of Columbia. Cancer Epidemiol Biomarkers Prev. 2012 Oct;21(10):1655-63. doi: 10.1158/1055-9965.EPI-12-0479. PMID 23045540
- [Background] Rabe F, Getachew S, Stroetmann CY, Mezger NCS, Gebremariam TY, Berhane B, Mremi A, Mmbaga BT, Boucheron P, McCormack V, Santos P, Addissie A, Kantelhardt EJ. Time to pathologic diagnosis of suspicious breast lesions: An institution-based study in five Ethiopian hospitals. Int J Cancer. 2025 Sep 1;157(5):876-889. doi: 10.1002/ijc.35436. Epub 2025 Apr 10. PMID 40207740
- [Background] Rohsig V, Silva P, Teixeira R, Lorenzini E, Maestri R, Saraiva T, Souza A. Nurse Navigation Program: Outcomes From a Breast Cancer Center in Brazil. Clin J Oncol Nurs. 2019 Feb 1;23(1):E25-E31. doi: 10.1188/19.CJON.E25-E31. PMID 30682003
- [Background] Khanna AS, Brickman B, Cronin M, Bergeron NQ, Scheel JR, Hibdon J, Calhoun EA, Watson KS, Strayhorn SM, Molina Y. Patient Navigation Can Improve Breast Cancer Outcomes among African American Women in Chicago: Insights from a Modeling Study. J Urban Health. 2022 Oct;99(5):813-828. doi: 10.1007/s11524-022-00669-9. Epub 2022 Aug 8. PMID 35941401
- [Background] Sankaranarayanan R, Ramadas K, Thara S, Muwonge R, Prabhakar J, Augustine P, Venugopal M, Anju G, Mathew BS. Clinical breast examination: preliminary results from a cluster randomized controlled trial in India. J Natl Cancer Inst. 2011 Oct 5;103(19):1476-80. doi: 10.1093/jnci/djr304. Epub 2011 Aug 23. PMID 21862730
- [Background] Provencher L, Hogue JC, Desbiens C, Poirier B, Poirier E, Boudreau D, Joyal M, Diorio C, Duchesne N, Chiquette J. Is clinical breast examination important for breast cancer detection? Curr Oncol. 2016 Aug;23(4):e332-9. doi: 10.3747/co.23.2881. Epub 2016 Aug 12. PMID 27536182
- [Background] Fuller MS, Lee CI, Elmore JG. Breast cancer screening: an evidence-based update. Med Clin North Am. 2015 May;99(3):451-68. doi: 10.1016/j.mcna.2015.01.002. Epub 2015 Mar 5. PMID 25841594
- [Background] Anderson BO, Ilbawi AM, Fidarova E, Weiderpass E, Stevens L, Abdel-Wahab M, Mikkelsen B. The Global Breast Cancer Initiative: a strategic collaboration to strengthen health care for non-communicable diseases. Lancet Oncol. 2021 May;22(5):578-581. doi: 10.1016/S1470-2045(21)00071-1. Epub 2021 Mar 7. No abstract available. PMID 33691141
- [Background] Dye TD, Bogale S, Hobden C, Tilahun Y, Hechter V, Deressa T, Bize M, Reeler A. Complex care systems in developing countries: breast cancer patient navigation in Ethiopia. Cancer. 2010 Feb 1;116(3):577-85. doi: 10.1002/cncr.24776. PMID 20029968
- [Background] Trabitzsch J, Wondimagegnehu A, Afework T, Stoeter O, Gizaw M, Getachew S, Feyisa JD, Taylor L, Wienke A, Addissie A, Kantelhardt EJ. Pathways and Referral of Patients with Cancer in Rural Ethiopia: A Multi-center Retrospective Cohort Study. Oncologist. 2023 Jun 2;28(6):e359-e368. doi: 10.1093/oncolo/oyad032. PMID 36940294
- [Background] Shita A, Yalew AW, Seife E, Afework T, Tesfaw A, Gufue ZH, Rabe F, Taylor L, Kantelhardt EJ, Getachew S. Survival and predictors of breast cancer mortality in South Ethiopia: A retrospective cohort study. PLoS One. 2023 Mar 6;18(3):e0282746. doi: 10.1371/journal.pone.0282746. eCollection 2023. PMID 36877683
- [Background] Tesfaw A, Getachew S, Addissie A, Jemal A, Wienke A, Taylor L, Kantelhardt EJ. Late-Stage Diagnosis and Associated Factors Among Breast Cancer Patients in South and Southwest Ethiopia: A Multicenter Study. Clin Breast Cancer. 2021 Feb;21(1):e112-e119. doi: 10.1016/j.clbc.2020.08.011. Epub 2020 Oct 1. PMID 33536135
- [Background] Joko-Fru WY, Miranda-Filho A, Soerjomataram I, Egue M, Akele-Akpo MT, N'da G, Assefa M, Buziba N, Korir A, Kamate B, Traore C, Manraj S, Lorenzoni C, Carrilho C, Hansen R, Finesse A, Somdyala N, Wabinga H, Chingonzoh T, Borok M, Chokunonga E, Liu B, Kantelhardt E, McGale P, Parkin DM. Breast cancer survival in sub-Saharan Africa by age, stage at diagnosis and human development index: A population-based registry study. Int J Cancer. 2020 Mar 1;146(5):1208-1218. doi: 10.1002/ijc.32406. Epub 2019 Jun 14. PMID 31087650
- [Background] Geremew H, Golla EB, Simegn MB, Abate A, Ali MA, Kumbi H, Wondie SG, Mengstie MA, Tilahun WM. Late-stage diagnosis: The driving force behind high breast cancer mortality in Ethiopia: A systematic review and meta-analysis. PLoS One. 2024 Jul 19;19(7):e0307283. doi: 10.1371/journal.pone.0307283. eCollection 2024. PMID 39028722
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751